CLINICAL TRIAL: NCT06781359
Title: An International Multicenter Observational Retrospective Study on Plasmablastic Lymphoma Patients
Brief Title: Study on Plasmablastic Lymphoma Patients
Acronym: FIL_PlaLy
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: AIL Roma - Italia (Unknown); AIL Cuneo - Italia (Unknown)
Responsible Party: Sponsor
Other Study IDs: FIL_PlaLy
Record Dates: First submitted 2024-12-05; First posted 2025-01-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Plasmablastic Lymphoma
Keywords: Plasmablastic lymphoma; PBL
MeSH Terms: conditions — Plasmablastic Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Histological and immunohistochemical slides used for the original diagnosis + block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Plasmablastic lymphoma patients: Patients with diagnosis (histologically confirmed) of plasmablastic lymphoma (PBL) between Jan 1st 2000 and Dec 31st 2022

SUMMARY:
This is an observational, multicenter, international and retrospective study, that aims to collect data on clinical and pathological characteristics, treatment regimens, outcome, and prognostic factors (clinical, biomarkers and/or radio-metabolic) in patients affected by PBL.

DETAILED DESCRIPTION:
This study is an International, multicenter, observational, retrospective trial on patients affected by PBL. The information collected aim to obtain data from the real-life diagnosis, staging, management and treatment and outcome of PBL patients. A centralized pathological review of pathological samples is planned to define the rate of accurate diagnosis and to define a recommended immunohistochemical diagnostic panel for PBL. In addition, exploratory analysis will be performed to better characterize PBL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plasmablastic lymphoma (PBL) between Jan 1st 2000, and Dec 31st 2022
* Histologically confirmed plasmablastic lymphoma (PBL) diagnosis according to local pathological report
* Age > 18 years old
* Availability of complete medical records
* Availability of histopathological material requested by the study

Exclusion Criteria:

* Any other histology than PBL
* Lack of complete medical records
* Lack of histopathological material requested by the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (Age ≥ 18 years old) with diagnosis of plasmablastic lymphoma (Histologically confirmed) between Jan 1st 2000, and Dec 31st 2022
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 36 months
  OS is defined as the time from the diagnosis to death for any cause or last clinical contact for censored patients.

SECONDARY OUTCOMES:
ECOG-PS | 36 months
  Proportion of Performance Status: from 0 (fully active) to 4 (Completely disabled)
Ann Arbor Stage | 36 months
  Proportion of stage: from I (better) to IV (worse)
Kidney and/or adrenal gland involvement | 36 months
  Proportion of the presence of involvement
Diagnostic liquor | 36 months
  Proportion of the presence of liquor
Splenic involvement | 36 months
  Proportion of spenic involvement
Type of chemotherapy (CHT) regimen | 36 months
  Proportion of CHT administered
Complete remission rate (CR) | 36 months
  CR at the end of treatment
Overall response rate (ORR) | 36 monts
  ORR is defined as the proportion of patients who have a partial or complete response to therapy
Progression-free survival (PFS) | 36 months
  PFS is defined as time from diagnosis to progression, relapse or death for any cause and last clinical contact for censored cases,
Validation of IPI and CNS-IPI score by means of Cox PH regression on OS and PFS | 36 months
  IPI (international prognostic Index) ranging from 0 (lower risk) to 5 points (greater risk); CNS-IPI score (Central Nervous System IPI) ranging from 0 (lower risk) to 6 points (greater risk).
Frequencies of HIV and EBV at relapse | 36 months
  Frequencies of HIV and EBV at relapse

CONTACTS AND LOCATIONS:
Overall Officials: Alessia Castellino, MD, Principal Investigator — UO Ematologia, AO Santa Croce e Carle, Cuneo - Italy; Emanuele Ravano, MD, Principal Investigator — UO Ematologia, Niguarda Grande Ospedale Metropolitano, Milano - Italy.
Locations (23):
- Italy (23):
  - IRCCS Centro di Riferimento Oncologico di Aviano, Divisione di Oncologia e dei Tumori immuno-correlati, Aviano, PN
  - Ospedale C.e G. Mazzoni, U.O.C. di Ematologia, Ascoli Piceno
  - ASST Spedali Civili di Brescia, Ematologia, Brescia
  - A.O. S. Croce e Carle, S.C. di Ematologia e Trapianto di Midollo Osseo, Cuneo
  - Azienda Ospedaliera Universitaria Careggi, Unità funzionale di Ematologia, Florence
  - ASST -Fatebenefratelli - Polo Luigi Sacco Oncologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, SC Ematologia, Milan
  - Istituto Scientifico San Raffaele, Unità Linfomi - Dipartimento Oncoematologia, Milan
  - Ospedale Maggiore Policlinico - Fondazione IRCCS Ca' Granda, Ematologia, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Ematologia, Monza
  - AOU Maggiore della Caritа di Novara, SCDU Ematologia, Novara
  - Azienda Ospedaliera Universitaria di Padova, Ematologia, Padua
  - Presidio ospedaliero A. Tortora, U.O. Onco-ematologia, Pagani
  - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Ematologia, Reggio Emilia
  - Azienda Ospedaliera Universitaria Sant' Andrea, Ematologia, Roma
  - Policlinico Umberto I - Università La Sapienza, Istituto Ematologia, Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - Universitа Cattolica S. Cuore, Ematologia, Roma
  - Azienda Ospedaliero Universitaria Senese, U.O.C. Ematologia, Siena
  - A.O.U. Città della Salute e della Scienza di Torino, Ematologia Universitaria, Torino
  - A.O.U. Città della Salute e della Scienza di Torino, S.C. Ematologia, Torino
  - Ospedale S. Chiara, S.S. di Ematologia, Trento
  - ULSS2 Marca Trevigiana, Ospedale Ca' Foncello, S.C di Ematologia, Treviso
  - ULSS 8 Berica - Ospedale S. Bortolo, Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may contact the FIL board at segreteriadirezione@filinf.it to share invidual-level patients' clinical data analysed for the publication article (for the avoidance of doubt, no identifiable data, such as name, address, hospital name, date of birth, or any other identifying data, will be shared and should not be requested).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: In compliance with the domestic ethics guideline and applicable legislation, invidual deindentified patients' data underlying the results reported in teh publication article (including study protocol, statistical analysis plan and data coding) can be shared until 5 years after the publication of the present article.
Access Criteria: For each data sharing request, it is essential that a proforma (available on request) is completed that describes the general purpose, specific aims, data items requested, analysis plan and acknowledgment of the trial management team. Requests will be reviewed based on scientific merit and ethical principles. Requestors who are granted access to the data will be required to complete a data sharing agreement that will be signed by the requester and FIL.